CLINICAL TRIAL: NCT00869882
Title: Comparison of 2 Surgical Approaches in the Treatment of Degenerative Spondylolysthesis: Posterolateral Fusion With Instrumentation (GPLI) Plus or Minus Transforaminal Lumbar Interbody Fusion (TLIF)
Brief Title: SPONGIT: Comparison of Two Surgical Approaches in the Treatment of Degenerative Spondylolysthesis
Acronym: SPONGIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2008/33
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Degenerative Spondylolisthesis
Keywords: Spondylolisthesis; degeneration; spinal fusion
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Posterolateral fusion with instrumentation combined to transforaminal lumbar interbody fusion
  Interventions: Procedure: Circumferential arthrodesis
- 2 (Active Comparator): Posterolateral fusion with instrumentation
  Interventions: Procedure: Posterolateral fusion with instrumentation

INTERVENTIONS:
Procedure: Circumferential arthrodesis — Patients are carefully positioned in the proned position and submitted to a posterior surgical approach under general anaesthesia. Surgical levels are viewed laterally by mean of intraoperative radiographs which can be performed at surgeon's demand during the whole surgery time.
  The preceding procedure is performed. In case of foraminal stenosis, decompression is performed at the same time as discal approach via the narrowest foramen.
  In addition to this, before preparation of bed for bone grafting, nerve roots are retracted and the disc nucleus is removed entirely, then endplate decortication is performed. The disc space is distracted. The most anterior part of the disc space is packed with cancellous bone. A cage packed with bone is inserted into the anterior portion of the interspace. According to cage location, bone graft could be inserted in the posterior portion of the interspace. Cage placement is radiologically checked.
  The end of the procedure is the same as for GPLI.
  Other Names: TLIF+GPLI
  Arms: 1
Procedure: Posterolateral fusion with instrumentation — Patients are carefully positioned in pronation and submitted to a posterior surgical approach under general anaesthesia. Surgical levels are viewed laterally by mean of intraoperative radiographs performed at surgeon's demand during the whole surgery time.
  Pedicle screw instrumentation is performed, followed by posterior neural decompression depending on the type of stenosis:
  * Central stenosis: decompression is performed including medial facectomy, laminectomy;
  * Foraminal stenosis: foraminotomy is performed, while preserving a graft bed as large as possible;
  * Pure foraminal stenosis: spinal duct is not opened. Local bone is harvested from the lamina and the spinous process and carefully fragmented for autologous graft.
  Subperiosteal dissection is performed between the transverse processes and lateral aspects of the facet joints.
  Two rods are placed and locked on screws in maximum compression to optimize segmental lordosis.
  Bone autograft is placed into this bed.
  Other Names: GPLI
  Arms: 2

SUMMARY:
This trial, conducted in adult patients with degenerative spondylolisthesis needing surgical treatment at one level, aimed at comparing two approaches of spinal fusion.

DETAILED DESCRIPTION:
Degenerative spondylolisthesis is defined as the slip of one vertebra onto the other due to degenerative lesions; the L4-L5 intervertebral space is mainly involved. Mean age of symptomatic disease is about 60. Surgery is indicated in the presence of radiculalgia and/or neurological claudication and/or invalidating lombalgia, worsening neurological deficit, presence of sphincterian incontinence.

Surgical treatment of degenerative spondylolisthesis usually consists in neural decompression followed by posterolateral fusion with instrumentation. In the literature, fusion rate is estimated to be 80% with GPLI and seems to be increased by interbody fusion, especially transforaminal lumbar interbody fusion which has the advantage of unilateral disc interspace route, and fusion rate over 90%.

It seems that hypolordosis in the instrumented segments caused increased loading of the posterior column in the adjacent segments. These biomechanical effects may explain the degenerative changes at the junction level that have been observed as long-term consequences of lumbar fusion.

In addition to fusion, segmental lordosis gain seems to be an important long-term prognostic factor. Segmental lordosis recovery (upper than 3° in order to take into account measurement variability), was never assessed after TLIF procedure nor compared to that after posterolateral fusion in controlled randomized clinical trials.

The main objective of the study is the comparison of efficacy between circumferential fusion (TLIF plus GPLI) and GPLI alone as surgical treatment of degenerative spondylolisthesis in term of "Success" rate, defined as fusion and at least 3-degree increase of segmental lordosis angle, 24 months after surgery.

In this trial, included patients will be randomly assigned to undergo either posterolateral fusion with instrumentation (GPLI) or circumferential fusion with transforaminal lumbar interbody fusion (TLIF) combined to GPLI. In both arms, bone autograft will be performed using loose fragments obtained during neurological decompression.

Six visits are planned during the study: pre-inclusion visit within 3 months before surgery, inclusion/randomisation on the day before surgery, 3 follow-up visits (2, 6, and 12 months after surgery) and an end of study visit 24 months after surgery (or at time of withdrawal if relevant). Hospital stay (about one week, on average) is planned after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged less than 75,
* Having been informed about clinical trial objectives and risk,
* Covered by health insurance system,
* Suffering from degenerative spondylolisthesis (whatever the grade and intervertebral disc height) needing one-level surgical fusion due to either invalidating lombalgia/radiculalgia despite 6-month optimal medical treatment and/or motor neurological symptoms.

Exclusion Criteria:

* Previous lumbar fusion,
* Previous spine traumatism,
* Presence of at least one major contraindication to surgery and/or general anaesthesia (ie, non controlled coagulopathy, active infection, or serious underlying disease, auto-immune affection).
* Presence of at least one contraindication to either TLIF or GPLI,
* Severe radiological osteoporosis.
* Active cancer at time of inclusion into the study.
* Unlikely to comply with the requirements of the study and/or to complete the study for psychological, social, familial or geographical reasons.
* Under any administrative or legal supervision.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Success rate defined as fusion associated to at least a 3-degree increase of segmental lordosis angle and the absence of a reintervention due to a failure of the initial intervention | 24 months after surgery

SECONDARY OUTCOMES:
Major complication (ie, life threatening haemorrhage, severe and persisting neurological worsening, deep infection) rate, and minor complication rate | within 24 months after surgery
Success rate defined as both fusion and at least 3-degree increase of segmental lordosis angle | 6 and 12 months after surgery
Lumbar and radicular pain outcome | 2, 6, 12 and 24 months after surgery
Functional outcome: Oswestry Disability Index and modified Prolo Economic and Functional scores | 2, 6, 12 and 24 months after surgery
Change of pelvic and radiological parameters (ie, lumbar lordosis angle, medial intervertebral space height | 2, 6, 12 and 24 months after surgery
Quality of life outcome: SF-36 | 2, 6, 12 and 24 months after surgery
Per and post operative surgery parameters (ie, operative time, blood loss, hospitalization stay duration) | within hospital stay due to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Patrick GUERIN, MD, Principal Investigator — University Hospital Bordeaux, France; Antoine BENARD, MD, Study Chair — University Hospital Bordeaux, France
Locations (1):
- Service de chirurgie orthopédique, Hôpital Pellegrin Tripode, Bordeaux, France

REFERENCES:
- [Background] Rosenberg NJ. Degenerative spondylolisthesis. Predisposing factors. J Bone Joint Surg Am. 1975 Jun;57(4):467-74. PMID 1141255
- [Background] Frymoyer JW. Degenerative Spondylolisthesis: Diagnosis and Treatment. J Am Acad Orthop Surg. 1994 Jan;2(1):9-15. doi: 10.5435/00124635-199401000-00002. PMID 10708989
- [Background] Cummins J, Lurie JD, Tosteson TD, Hanscom B, Abdu WA, Birkmeyer NJ, Herkowitz H, Weinstein J. Descriptive epidemiology and prior healthcare utilization of patients in the Spine Patient Outcomes Research Trial's (SPORT) three observational cohorts: disc herniation, spinal stenosis, and degenerative spondylolisthesis. Spine (Phila Pa 1976). 2006 Apr 1;31(7):806-14. doi: 10.1097/01.brs.0000207473.09030.0d. PMID 16582855
- [Background] Taylor VM, Deyo RA, Cherkin DC, Kreuter W. Low back pain hospitalization. Recent United States trends and regional variations. Spine (Phila Pa 1976). 1994 Jun 1;19(11):1207-12; discussion 13. doi: 10.1097/00007632-199405310-00002. PMID 8073311
- [Background] Brown MD, Lockwood JM. Degenerative spondylolisthesis. Instr Course Lect. 1983;32:162-9. PMID 6546064
- [Background] Kostuik JP, Harrington I, Alexander D, Rand W, Evans D. Cauda equina syndrome and lumbar disc herniation. J Bone Joint Surg Am. 1986 Mar;68(3):386-91. PMID 2936744
- [Background] Magora A. Conservative treatment in spondylolisthesis. Clin Orthop Relat Res. 1976 Jun;(117):74-9. PMID 132329
- [Background] Matsunaga S, Ijiri K, Hayashi K. Nonsurgically managed patients with degenerative spondylolisthesis: a 10- to 18-year follow-up study. J Neurosurg. 2000 Oct;93(2 Suppl):194-8. doi: 10.3171/spi.2000.93.2.0194. PMID 11012048
- [Background] Herkowitz HN. Spine update. Degenerative lumbar spondylolisthesis. Spine (Phila Pa 1976). 1995 May 1;20(9):1084-90. doi: 10.1097/00007632-199505000-00018. PMID 7631240
- [Background] Weinstein JN, Tosteson TD, Lurie JD, Tosteson AN, Blood E, Hanscom B, Herkowitz H, Cammisa F, Albert T, Boden SD, Hilibrand A, Goldberg H, Berven S, An H; SPORT Investigators. Surgical versus nonsurgical therapy for lumbar spinal stenosis. N Engl J Med. 2008 Feb 21;358(8):794-810. doi: 10.1056/NEJMoa0707136. PMID 18287602
- [Background] Atlas SJ, Keller RB, Robson D, Deyo RA, Singer DE. Surgical and nonsurgical management of lumbar spinal stenosis: four-year outcomes from the maine lumbar spine study. Spine (Phila Pa 1976). 2000 Mar 1;25(5):556-62. doi: 10.1097/00007632-200003010-00005. PMID 10749631
- [Background] Herkowitz HN, Kurz LT. Degenerative lumbar spondylolisthesis with spinal stenosis. A prospective study comparing decompression with decompression and intertransverse process arthrodesis. J Bone Joint Surg Am. 1991 Jul;73(6):802-8. PMID 2071615
- [Background] Gibson JN, Grant IC, Waddell G. The Cochrane review of surgery for lumbar disc prolapse and degenerative lumbar spondylosis. Spine (Phila Pa 1976). 1999 Sep 1;24(17):1820-32. doi: 10.1097/00007632-199909010-00012. PMID 10488513
- [Background] Fischgrund JS, Mackay M, Herkowitz HN, Brower R, Montgomery DM, Kurz LT. 1997 Volvo Award winner in clinical studies. Degenerative lumbar spondylolisthesis with spinal stenosis: a prospective, randomized study comparing decompressive laminectomy and arthrodesis with and without spinal instrumentation. Spine (Phila Pa 1976). 1997 Dec 15;22(24):2807-12. doi: 10.1097/00007632-199712150-00003. PMID 9431616
- [Background] Kornblum MB, Fischgrund JS, Herkowitz HN, Abraham DA, Berkower DL, Ditkoff JS. Degenerative lumbar spondylolisthesis with spinal stenosis: a prospective long-term study comparing fusion and pseudarthrosis. Spine (Phila Pa 1976). 2004 Apr 1;29(7):726-33; discussion 733-4. doi: 10.1097/01.brs.0000119398.22620.92. PMID 15087793
- [Background] Bono CM, Lee CK. Critical analysis of trends in fusion for degenerative disc disease over the past 20 years: influence of technique on fusion rate and clinical outcome. Spine (Phila Pa 1976). 2004 Feb 15;29(4):455-63; discussion Z5. doi: 10.1097/01.brs.0000090825.94611.28. PMID 15094543
- [Background] Ray CD. Threaded titanium cages for lumbar interbody fusions. Spine (Phila Pa 1976). 1997 Mar 15;22(6):667-79; discussion 679-80. doi: 10.1097/00007632-199703150-00019. PMID 9089940
- [Background] Ekman P, Moller H, Tullberg T, Neumann P, Hedlund R. Posterior lumbar interbody fusion versus posterolateral fusion in adult isthmic spondylolisthesis. Spine (Phila Pa 1976). 2007 Sep 15;32(20):2178-83. doi: 10.1097/BRS.0b013e31814b1bd8. PMID 17873808
- [Background] Kim KT, Lee SH, Lee YH, Bae SC, Suk KS. Clinical outcomes of 3 fusion methods through the posterior approach in the lumbar spine. Spine (Phila Pa 1976). 2006 May 20;31(12):1351-7; discussion 1358. doi: 10.1097/01.brs.0000218635.14571.55. PMID 16721298
- [Background] Dantas FL, Prandini MN, Ferreira MA. Comparison between posterior lumbar fusion with pedicle screws and posterior lumbar interbody fusion with pedicle screws in adult spondylolisthesis. Arq Neuropsiquiatr. 2007 Sep;65(3B):764-70. doi: 10.1590/s0004-282x2007000500006. PMID 17952277
- [Background] La Rosa G, Cacciola F, Conti A, Cardali S, La Torre D, Gambadauro NM, Tomasello F. Posterior fusion compared with posterior interbody fusion in segmental spinal fixation for adult spondylolisthesis. Neurosurg Focus. 2001 Apr 15;10(4):E9. doi: 10.3171/foc.2001.10.4.10. PMID 16732636
- [Background] Humphreys SC, Hodges SD, Patwardhan AG, Eck JC, Murphy RB, Covington LA. Comparison of posterior and transforaminal approaches to lumbar interbody fusion. Spine (Phila Pa 1976). 2001 Mar 1;26(5):567-71. doi: 10.1097/00007632-200103010-00023. PMID 11242386
- [Background] Hackenberg L, Halm H, Bullmann V, Vieth V, Schneider M, Liljenqvist U. Transforaminal lumbar interbody fusion: a safe technique with satisfactory three to five year results. Eur Spine J. 2005 Aug;14(6):551-8. doi: 10.1007/s00586-004-0830-1. Epub 2005 Jan 26. PMID 15672243
- [Background] Hee HT, Castro FP Jr, Majd ME, Holt RT, Myers L. Anterior/posterior lumbar fusion versus transforaminal lumbar interbody fusion: analysis of complications and predictive factors. J Spinal Disord. 2001 Dec;14(6):533-40. doi: 10.1097/00002517-200112000-00013. PMID 11723406
- [Background] Lauber S, Schulte TL, Liljenqvist U, Halm H, Hackenberg L. Clinical and radiologic 2-4-year results of transforaminal lumbar interbody fusion in degenerative and isthmic spondylolisthesis grades 1 and 2. Spine (Phila Pa 1976). 2006 Jul 1;31(15):1693-8. doi: 10.1097/01.brs.0000224530.08481.4e. PMID 16816765
- [Background] Lowe TG, Tahernia AD. Unilateral transforaminal posterior lumbar interbody fusion. Clin Orthop Relat Res. 2002 Jan;(394):64-72. doi: 10.1097/00003086-200201000-00008. PMID 11795753
- [Background] McAfee PC, DeVine JG, Chaput CD, Prybis BG, Fedder IL, Cunningham BW, Farrell DJ, Hess SJ, Vigna FE. The indications for interbody fusion cages in the treatment of spondylolisthesis: analysis of 120 cases. Spine (Phila Pa 1976). 2005 Mar 15;30(6 Suppl):S60-5. doi: 10.1097/01.brs.0000155578.62680.dd. PMID 15767888
- [Background] Potter BK, Freedman BA, Verwiebe EG, Hall JM, Polly DW Jr, Kuklo TR. Transforaminal lumbar interbody fusion: clinical and radiographic results and complications in 100 consecutive patients. J Spinal Disord Tech. 2005 Aug;18(4):337-46. doi: 10.1097/01.bsd.0000166642.69189.45. PMID 16021015
- [Background] Salehi SA, Tawk R, Ganju A, LaMarca F, Liu JC, Ondra SL. Transforaminal lumbar interbody fusion: surgical technique and results in 24 patients. Neurosurgery. 2004 Feb;54(2):368-74; discussion 374. doi: 10.1227/01.neu.0000103493.25162.18. PMID 14744283
- [Background] Umehara S, Zindrick MR, Patwardhan AG, Havey RM, Vrbos LA, Knight GW, Miyano S, Kirincic M, Kaneda K, Lorenz MA. The biomechanical effect of postoperative hypolordosis in instrumented lumbar fusion on instrumented and adjacent spinal segments. Spine (Phila Pa 1976). 2000 Jul 1;25(13):1617-24. doi: 10.1097/00007632-200007010-00004. PMID 10870136
- [Background] Kumar MN, Baklanov A, Chopin D. Correlation between sagittal plane changes and adjacent segment degeneration following lumbar spine fusion. Eur Spine J. 2001 Aug;10(4):314-9. doi: 10.1007/s005860000239. PMID 11563617
- [Background] Champain S, Benchikh K, Nogier A, Mazel C, Guise JD, Skalli W. Validation of new clinical quantitative analysis software applicable in spine orthopaedic studies. Eur Spine J. 2006 Jun;15(6):982-91. doi: 10.1007/s00586-005-0927-1. Epub 2005 Jun 17. PMID 15965708
- [Background] Bridwell KH, Lenke LG, McEnery KW, Baldus C, Blanke K. Anterior fresh frozen structural allografts in the thoracic and lumbar spine. Do they work if combined with posterior fusion and instrumentation in adult patients with kyphosis or anterior column defects? Spine (Phila Pa 1976). 1995 Jun 15;20(12):1410-8. PMID 7676341
- [Background] Rillardon L, Levassor N, Guigui P, Wodecki P, Cardinne L, Templier A, Skalli W. [Validation of a tool to measure pelvic and spinal parameters of sagittal balance]. Rev Chir Orthop Reparatrice Appar Mot. 2003 May;89(3):218-27. French. PMID 12844045
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Prolo DJ, Oklund SA, Butcher M. Toward uniformity in evaluating results of lumbar spine operations. A paradigm applied to posterior lumbar interbody fusions. Spine (Phila Pa 1976). 1986 Jul-Aug;11(6):601-6. doi: 10.1097/00007632-198607000-00012. PMID 3787326
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Finlay AY. Quality of life assessments in dermatology. Semin Cutan Med Surg. 1998 Dec;17(4):291-6. doi: 10.1016/s1085-5629(98)80026-6. PMID 9859917